CLINICAL TRIAL: NCT05372523
Title: Pilot Investigation of Senseye's Ocular Brain-Computer Interface (OBCI) for Diagnosis of Adult With Post-Traumatic Stress Disorder (PTSD)
Brief Title: Senseye's OBCI Diagnostic Tool for PTSD
Status: Terminated | Type: Observational
Why Stopped: No participants completed study
Sponsor: Senseye, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SEN-01-2022
Record Dates: First submitted 2022-04-27; First posted 2022-05-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Trauma+ & PTSD: Patients diagnosed with significant trauma exposure and PTSD
  Interventions: Diagnostic Test: CAPS-5 Assessment; Diagnostic Test: Senseye OBCI
- Trauma+ & No PTSD: Patients diagnosed with significant trauma exposure but no PTSD
  Interventions: Diagnostic Test: CAPS-5 Assessment; Diagnostic Test: Senseye OBCI
- No trauma or PTSD: Healthy adults without known major psychiatric disorders
  Interventions: Diagnostic Test: CAPS-5 Assessment; Diagnostic Test: Senseye OBCI

INTERVENTIONS:
Diagnostic Test: CAPS-5 Assessment — A validated, semi-structured clinical interview to assess core PTSD symptoms
Diagnostic Test: Senseye OBCI — Using a machine learning algorithm, Senseye's DT will record a series of visual tasks, pupil light reflex, vascular function and heart rate measurement throughout.

SUMMARY:
This pilot study will investigate the feasibility, acceptability, repeatability, accuracy and efficacy of the Senseye OBCI diagnostic tool to assess the presence and severity of PTSD symptoms and monitor response to trauma-informed interventions. A total of 68 adults will be included in the study with a follow-up time point of 9 weeks post-initial intervention.

DETAILED DESCRIPTION:
This pilot study will investigate the feasibility, acceptability, repeatability, accuracy, and efficacy of operator-independent Senseye Ocular Brain-Computer Interface (OBCI) diagnostic tool to assess the presence and severity of PTSD symptoms and monitor response to trauma-informed interventions. After informed consent, 68 adults - 34 with PTSD and 17 adults with significant trauma exposure but no PTSD, and 17 healthy adults without known major psychiatric disorders, aged 18-65 years old, will be recruited and undergo OBCI diagnostic tool, comparing against gold standards tools- the CAPS-5, UCLA PTSD Reaction Index for DSM-5 (PTSD-RI). Fifteen participants will undergo repeatability and reproducibility assessments. Adults with PTSD will receive a standard of care trauma-informed interventions for eight weeks, and their biopsychosocial characteristics, Senseye OBCI, neuropsychiatric measures will be measured at baseline and week 9. Using Senseye's machine learning algorithm, Senseye OBCI will use a facecam recorder during a series of visual tasks, pupil light reflex, and heart rate measurement throughout.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female diagnosed with PTSD (only for PTSD group)
2. aged 18- 65 years old
3. able to read/write in English

Exclusion Criteria:

1. presence of intellectual disabilities
2. psychotic or self-injurious behavior
3. seizure disorder
4. major depression
5. traumatic brain injury (TBI)
6. language disorder
7. eye disorders
8. other neurodevelopmental disorders
9. history of lifetime psychosis
10. mania
11. current suicidality
12. diagnosis of a substance use disorder
13. impaired functioning to the degree that requires immediate initiation of psychotropic medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults presenting to the clinic with potential psychiatric disorder, to include PTSD
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Agreement between Senseye OBCI measures and gold-standard measures | 9 weeks
  Assessments for the presence and severity of PTSD symptoms will be compared between the Senseye tool and the gold-standard measures for percent agreement.
Feasibility of the Senseye tool | 9 weeks
  Feasibility will be assessed by evaluating retention rate.
Test-retest for repeatability of the Senseye tool | 1 week
  Senseye OBCI assessments will be repeated the same day and again at one week.

SECONDARY OUTCOMES:
Prognostic value by comparing Senseye OBCI to core PTSD symptoms | 9 weeks
  Analyses of data collected on the Senseye tool will be compared with the core PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Naser Ahmadi, MD, Principal Investigator — Olive View - UCLA
Locations (1):
- Olive View - UCLA Medical Center, Sylmar, California, United States